CLINICAL TRIAL: NCT04129359
Title: FamilieTrivsel i Almen Praksis: A General Practice-based Cluster-randomised Trial of the Impact of the Resilience Programme on Early Child Development
Brief Title: FamilieTrivsel i Almen Praksis: a Mentalisation Programme for Families With Young Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Research Unit Of General Practice, Copenhagen (Other)
Collaborators: TrygFonden, Denmark (Industry); Göteborg University (Other); University of Aberdeen (Other); University of Southern Denmark (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jakob Kragstrup, Professor of General Practice, Research Unit Of General Practice, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0001
Record Dates: First submitted 2019-10-08; First posted 2019-10-16 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Parent-Child Relations; Child Development; Parenting

STUDY DESIGN:
Intervention Model Description: Cluster RCT in general practices, which will recruit successive pregnant women. All practices will receive training in data recording and assessment, and half will receive additional training in use of the online intervention. Our original sample size calculation required 1,000 participants, in 100 clusters of 10 participants per practice. This would allow us to detect a difference of two points in the SDQ Total Difficulties Scale score (an effect size of 0.3) with 90% power at a 2.5% significance level assuming the intraclass correlation coefficient was 0.06. We continued to recruit practices until COVID-19 restrictions prevented further recruitment of practices. We then made a decision to increase the cluster size, allowing participating practices to recruit up to 30 participants. We were also able to adjust our original estimate of the intra-class correlation coefficient based on our baseline data from 0.06 to 0.02 allowing us to reduce our target sample size from 1000 to 624.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FamilieTrivsel (Experimental): Enhanced care as usual in general practice plus training in the use of the online mentalisation programme
  Interventions: Behavioral: FamilieTrivsel; Other: enhanced care as usual
- control (Active Comparator): Enhanced care as usual in general practice
  Interventions: Other: enhanced care as usual

INTERVENTIONS:
Behavioral: FamilieTrivsel — FamilieTrivsel is a modular internet-based low-cost and brief psychoeducation intervention based on the Robusthed (Resilience) programme (RP). Mentalisation approaches are used to increase resilience and ability to handle the challenges of life. The programme is licence free and can be used with low or high intensity and it can be combined with any other interventions. RP provides simple explanations and tools that can be used to discover, understand and regulate one's own thoughts and feelings by activating mental and physical resources and it provides examples and exercises that may promote communication about mental states between parents and the child. The content has been developed to include video-based training sessions based on different stages of pregnancy and early childrearing. RP appears suitable for use in general practice, where the GP sees young parents regularly and thus can direct patients towards components of the programme when need appears greatest.
  Other Names: Robustbarn.dk (FamilieTrivsel is a customised variant focused on families with young children)
  Arms: FamilieTrivsel
Other: enhanced care as usual — Structured assessments of maternal mental health, child neurodevelopment and parent-child interaction in routine preventive health care in general practice
  Other Names: control

SUMMARY:
This cluster randomised trial aims to establish the effectiveness of an online intervention designed to improve the ability of parents to 'mentalise' - in other words to understand their own mental states and that of others including their partners and young children. Effects on maternal mental state, the quality of parent-child interaction and child language, social and emotional development will be assessed.

DETAILED DESCRIPTION:
This is a cluster randomised trial based in Danish general practice. A number of general practitioners will be recruited, each of which will recruit successive women at their first routine antenatal appointment. All practices will receive standardised training in assessing maternal mental health, neurodevelopmental assessment of the child and assessment of the quality of parent-child interaction as well as in completion of an enhanced pregnancy or child development record.

Practices will be randomised either to receive additional training in the principles of mentalisation and in the use of an online resource (Robusthed) that parents can use to improve their mentalisation skills (https://robustbarn.dk) or not to receive this extra training. The trial is therefore comparing Robusthed plus enhanced care as usual with enhanced care as usual alone.

Baseline measures will be taken at recruitment into the trial and outcomes will be collected when the child is 15 and 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women presenting at their first GP-based antenatal assessment and their families

Exclusion Criteria:

* Non-Danish speaking women
* Families planning to move to a new general practice during the pregnancy or shortly after the birth of the child
* Mother has already participated in the trial (e.g., second eligible baby within life of the study)
* Presentation to the GP after the time for the third scheduled antenatal visit
* Miscarriage or other pregnancy loss after recruitment to the study will lead to late exclusion from the study
* Second pregnancies among already-participating families

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 624 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire Total Difficulties Score | 30 months postnatal
  Child psychiatric symptom score, range from 0-40, parent complete, lower scores indicate better outcome.
MacArthur-Bates Communicative Development Inventory (100 word Danish version) | 30 months postnatal
  Child expressive language measure - range 0-100 - parent complete - higher scores indicate better outcomes

SECONDARY OUTCOMES:
Child-Adult Relationship Observation (CARO) | 30 months post natal
  Event-based scoring system counting rates of positive and negative parenting behaviours in a home-based video of a caring episode (eg mealtime). Blinded rater. Positive and negative scores 0-6, high positive scores and low negative scores are better outcomes.
Hospital Anxiety and Depression Scale | 30 months postnatal
  Scores for anxiety and depression (parent self-complete) - separate scores for anxiety and depression - both scales range 0-21 - on both scales low scores indicate better outcome
Service and societal costs | 30 months postnatal
  Within-trial costs of participants' service use and out of pocket expenses - collected by parental questionnaire
EQ-5D-5L (EuroQol 5-Dimension 5-Level) | 30 months postnatal
  Maternal health-related quality of life - parental self-complete - range 5-25 - low scores indicate better outcome
EQ VAS (EuroQol Visual Analog Scale) | 30 months postnatal
  Maternal self rated health - range 0-100 - high scores indicate better outcome.

OTHER OUTCOMES:
Child-Adult Relationship Observation (CARO) | 15 months postnatal
  Event-based scoring system counting rates of positive and negative parenting behaviours in a home-based video of a caring episode (eg mealtime). Blinded rater. Positive and negative scores 0-6, high positive scores and low negative scores are better outcomes.
Maternal Hospital Anxiety and Depression Scale | 15 months postnatal
  separate scores for anxiety and depression (parent self-complete) - both scales range 0-21 - on both scales low scores indicate better outcome
Service and societal costs | 15 months postnatal
  Within-trial costs of participants' service use and out of pocket expenses - collected by parental questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philip Wilson, DPhil FRCGP, Principal Investigator — University of Copenhagen
Locations (1):
- Capital Region, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
To be determined
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Protocol to be published during recruitment phase. SAP to be published before unblinding.
Access Criteria: Open access once published

REFERENCES:
- [Derived] Stroyer de Voss S, Wilson PMJ, Kirk Ertmann R, Overbeck G. Increased family psychosocial focus during children's developmental assessments: a study of parents' views. BMC Pediatr. 2024 May 15;24(1):335. doi: 10.1186/s12887-024-04800-4. PMID 38750557
- [Derived] Sorensen ER, Rasmussen IS, Overbeck G, Siersma V, Appel CL, Wilson P. Uptake of signposting to web-based resources: pregnant women's use of a preventive web-based intervention. BMC Prim Care. 2023 Sep 16;24(1):189. doi: 10.1186/s12875-023-02130-5. PMID 37716967
- [Derived] de Voss S, Wilson P, Saxild S, Overbeck G. Increasing the psychosocial focus in child developmental assessments: a qualitative study. BMC Pediatr. 2023 Jan 25;23(1):44. doi: 10.1186/s12887-023-03849-x. PMID 36698093
- [Derived] Overbeck G, Kragstrup J, Gortz M, Rasmussen IS, Graungaard AH, Siersma V, de Voss S, Ertmann RK, Shahrzad S, Appel CL, Wilson P. Family wellbeing in general practice: a study protocol for a cluster-randomised trial of the web-based resilience programme on early child development. Trials. 2023 Jan 4;24(1):7. doi: 10.1186/s13063-022-07045-7. PMID 36597136